CLINICAL TRIAL: NCT05005130
Title: Mixed Methods Formative Research and Pilot Testing of a Task-shifted Adaptation of the WHO-PEN Intervention to Address Cardio-metabolic Complications in People Living With HIV in Zambia
Brief Title: Task-shifted Adaptation of the WHO-PEN Intervention to Address Cardio-metabolic Complications in People Living With HIV in Zambia
Acronym: TASKPEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Centre for Infectious Disease Research in Zambia (Other); University of Zambia (Other); Ministry of Health, Zambia (Other Government); University of Alabama at Birmingham (Other); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 20-3606; UG3HL156389 (NIH)
Record Dates: First submitted 2021-07-19; First posted 2021-08-13 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2023-11

CONDITIONS: Non Communicable Diseases; HIV
Keywords: HIV; Non Communicable Diseases; WHO-PEN
MeSH Terms: conditions — Noncommunicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cluster 1 (George) (Experimental): 3 months without TASKPEN (Standard of Care) and 6 months with TASKPEN.
  Interventions: Other: TASKPEN
- Cluster 2 (Chilengi) (Experimental): 6 months without TASKPEN (Standard of Care) and 3 months with TASKPEN
  Interventions: Other: TASKPEN

INTERVENTIONS:
Other: TASKPEN — TASKPEN is the name of the package of implementation strategies proposed by the investigators that are intended to deliver the WHO PEN intervention in routine HIV clinical practice settings in Zambia. TASKPEN has five components which will be the subject of stakeholder consultation and adaptation in this formative research protocol. The package of integrated HIV/NCD services includes:
  1. WHO PEN protocols, algorithm, & training materials adapted for Zambia
  2. Access to cardio-metabolic condition screening & laboratory monitoring
  3. Non communicable disease-focused electronic medical record module
  4. Integrated non-communicable/HIV care ("one stop shop" for services)
  5. Strengthened non-communicable disease (NCD) medication supply chain, including multi-month dispensing (MMD)

SUMMARY:
This mixed-methods formative research study aims to adapt the WHO Package of Essential Noncommunicable Disease Interventions (WHO-PEN) approach for the Zambian public health system, and pilot test an adapted, streamlined, and task-shifted package of integrated HIV Noncommunicable Disease (NCD) services, collectively called "TASKPEN".

DETAILED DESCRIPTION:
Using local data and implementation science theories WHO-PEN will be adapted for Zambia, and TASKPEN developed to focus on addressing challenges faced by persons living with HIV (PLHIV) who have cardio-metabolic complications related to HIV or its treatment (e.g. hypertension, diabetes, dyslipidaemia). TASKPEN aims to improve detection and management of these complications.

Formative research activities for objective 1 include focus group discussions (FGDs), surveys and interviews with key stakeholders, which will include in-depth interviews (IDIs) with patients.

Objective 2 launches the TASKPEN pilot and fully task-shifts the TASKPEN package to non-physician healthcare workers (NPHWs) and integrates it within the President's Emergency Plan for AIDS Relief (PEPFAR) -supported HIV service delivery platform. A mix of IDIs, FGDs, key informant interviews, and patient and implementation surveys with implementation actors to evaluate feasibility, acceptability, and other implementation outcomes

ELIGIBILITY:
Objective 1

Focus group discussion participants/implementation survey participants:

Inclusion:

* 18 years of age or older
* non-physician professional or lay/peer health care worker (HCW) involved with HIV and/or NCD service delivery.

Key Informant Interview (KII) participants:

* 18 years of age or older
* a senior Ministry of Health (MOH) policy maker or health official working at national level in Zambia involved in managing, coordinating, and/or overseeing health services for non-communicable diseases in Zambia.

In-depth interview participants:

* emancipated HIV-infected adults 18 years of age or older have a documented cardio-metabolic condition

Exclusion:

* any potential IDI, FGD, or KII participant if they are unwilling or unable to provide informed consent.

Objective 2:

Cross-sectional assessments:

Inclusion:

* HIV-infected
* aged 18 years and older
* seeking care at either of the two ACHIEVE-supported pilot sites who are screened for and/or found to have evidence of one or more of the cardio-metabolic conditions or risk factors.

Nested cohort participants:

Inclusion:

* documented HIV infection
* aged 18 years or older
* have one or more cardio-metabolic conditions or risk factors:

  * obesity (defined as BMI > 30 kg/m^2);
  * any current tobacco smoking;
  * hypertension as defined by WHO PEN (i.e., systolic blood pressure (SBP) = 140 mmHg and/or diastolic blood pressure (DBP) = 90 mmHg);
  * diabetes mellitus as defined by WHO PEN (i.e. random plasma glucose = 11.1 mmol/L, fasting plasma glucose = 7 mmol/L, and/or haemoglobin A1c = 48 mmol/mol);
  * prediabetes (defined as having impaired fasting glucose of 6.1 to 6.9 mmol/L, impaired glucose tolerance with a two-hour, post-oral glucose tolerance test glucose =7.8 mmol/L but <11.1 mmol/L and a fasting plasma glucose <7.0 mmol/L, and/or haemoglobin A1c 42 to 48 mmol/mol); 6) dyslipidaemia (defined as total cholesterol >4 mmol/L or low density lipoprotein =6 mmol/L); and/or 7) personal history or medication use for heart disease, heart failure, stroke, or other cardio-metabolic complication (including but not limited to coronary artery disease, cerebrovascular disease, myocardial infarction, stroke, or peripheral vascular disease).

IDI participants:

* HIV-infected
* 18 years of age who were enrolled in the nested cohort and had documented exposure to the TASKPEN intervention at a pilot site.

FGD participants:

* 18 years of age or older
* a non physician health care worker (NPHW) or community health worker (CHW)/ lay health provider involved with TASKPEN or integrated HIV/NCD service delivery generally familiar with HIV and/or NCD service delivery at their facility.

KII participants:

* 18 years of age or older
* a facility-level antiretroviral therapy (ART) or out-patient department (OPD) clinic manager/ in-charge or policy maker at district, provincial, or national level in Zambia; and generally familiar with HIV and/or NCD-related issues in their community.

Exclusion criteria:

For the nested cohort component, investigators will exclude:

* adults who have no documented evidence of having established HIV care at the sites.
* people unlikely to remain at the site to the completion of the study follow-up.
* any potential IDI, FGD, or KII participant if they are unwilling or unable to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1129 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Herce, MD, MPH, MSc, Principal Investigator — University of North Carolina; Wilbroad Mutale, MBChB, MPhil, MPhil, PhD, Principal Investigator — Centre for Infectious Disease Research in Zambia
Locations (4):
- Zambia (4):
  - Chawama 1st Level hospital, Lusaka
  - Chilenje 1st level hospital, Lusaka
  - George urban health center, Lusaka
  - Mtendere health center, Lusaka

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC
Time Frame: from 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 28 Healthcare Providers and 1101 patient participants were enrolled and 11 were excluded from the analysis. This 'mini' stepped wedge pilot had 2 clinic clusters to establish approach feasibility. In a stepped wedge fashion, participants at both clinics were surveyed at baseline and then one site was randomly selected to receive the intervention for 3 months. A midline survey was then conducted and the second site was switched to the intervention before an endline survey 3 months later.
Units Other Than Participants: Clinics
Groups:
- Cluster 1 (George): 3 months without TASKPEN (Standard of Care (SOC)) and 6 months with TASKPEN.
  During the control period, participants receive the current standard of care (SOC) in Zambia. Under the SOC in Zambian health facilities, the screening, diagnosis, and treatment of cardio-metabolic NCDs are generally unavailable in the clinical departments where most PLHIV seek and receive health services (i.e., ART and DSD clinics), and typically are only offered for hypertension in the general outpatient medical settings that provide urgent care-like services. Under the SOC, health worker capacity to diagnose and manage cardio-metabolic NCDs, including among non-physicians and community health workers, is severely limited and not protocolized like HIV services.
  During the intervention period, participants receive TASKPEN package of integrated HIV/NCD services:
  1. WHO PEN protocols, algorithm, & training materials adapted for Zambia
  2. Access to cardio-metabolic condition screening & laboratory monitoring
  3. Non communicable disease-focused electronic medical record module
  4. Integrated non-communicable/HIV care ("one stop shop" for services)
  5. Strengthened non-communicable disease (NCD) medication supply chain, including multi-month dispensing (MMD).
- Cluster 2 (Chilenje): 6 months without TASKPEN (Standard of Care (SOC)) and 3 months with TASKPEN
  During the control period, participants receive the current standard of care (SOC) in Zambia. Under the SOC in Zambian health facilities, the screening, diagnosis, and treatment of cardio-metabolic NCDs are generally unavailable in the clinical departments where most PLHIV seek and receive health services (i.e., ART and DSD clinics), and typically are only offered for hypertension in the general outpatient medical settings that provide urgent care-like services. Under the SOC, health worker capacity to diagnose and manage cardio-metabolic NCDs, including among non-physicians and community health workers, is severely limited and not protocolized like HIV services.
  During the intervention period, participants receive TASKPEN package of integrated HIV/NCD services:
  1. WHO PEN protocols, algorithm, & training materials adapted for Zambia
  2. Access to cardio-metabolic condition screening & laboratory monitoring
  3. Non communicable disease-focused electronic medical record module
  4. Integrated non-communicable/HIV care ("one stop shop" for services)
  5. Strengthened non-communicable disease (NCD) medication supply chain, including multi-month dispensing (MMD).
Period: Time Period 1 Baseline (T0)
Arm/Group | Cluster 1 (George) | Cluster 2 (Chilenje)
Started (Unique patient participants enrolled into each Time Period.) | 227; 1 Clinics (SOC Control) | 221; 1 Clinics (SOC Control)
Healthcare Providers | 20; 1 Clinics | 0; 0 Clinics
Completed | 226; 1 Clinics | 221; 1 Clinics
Not Completed | 1; 0 Clinics | 0; 0 Clinics
Period: Time Period 2 Midline Survey (T1)
Arm/Group | Cluster 1 (George) | Cluster 2 (Chilenje)
Started (Unique patient participants enrolled into each time period.) | 188; 1 Clinics (TASKPEN Intervention) | 188; 1 Clinics (SOC Control)
Completed | 187; 1 Clinics | 186; 1 Clinics
Not Completed | 1; 0 Clinics | 2; 0 Clinics
Period: Time Period 3 Endline Survey (T2)
Arm/Group | Cluster 1 (George) | Cluster 2 (Chilenje)
Started (Unique patient participants enrolled into each time period.) | 158; 1 Clinics (TASKPEN Intervention) | 119; 1 Clinics (TASKPEN Intervention)
Healthcare Providers | 0; 0 Clinics | 8; 1 Clinics
Completed | 152; 1 Clinics | 118; 1 Clinics
Not Completed | 6; 0 Clinics | 1; 0 Clinics

BASELINE CHARACTERISTICS:
Population: Data are reported for those patient participants who had complete primary outcomes.
Groups:
- Standard of Care Patients: During the control period, participants receive the current standard of care (SOC) in Zambia. Under the SOC in Zambian health facilities, the screening, diagnosis, and treatment of cardio-metabolic NCDs are generally unavailable in the clinical departments where most PLHIV seek and receive health services (i.e., ART and DSD clinics), and typically are only offered for hypertension in the general outpatient medical settings that provide urgent care-like services. Under the SOC, health worker capacity to diagnose and manage cardio-metabolic NCDs, including among non-physicians and community health workers, is severely limited and not protocolized like HIV services.
- TASKPEN Patients: During the intervention period, participants receive TASKPEN intervention services.
  TASKPEN: The package of integrated HIV/NCD services:
  1. WHO PEN protocols, algorithm, & training materials adapted for Zambia
  2. Access to cardio-metabolic condition screening & laboratory monitoring
  3. Non communicable disease-focused electronic medical record module
  4. Integrated non-communicable/HIV care ("one stop shop" for services)
  5. Strengthened non-communicable disease (NCD) medication supply chain, including multi-month dispensing (MMD)
- Standard of Care Healthcare Providers; TASKPEN Healthcare Providers: Healthcare Providers employed at either of the clinics who participated in study surverys.
- Total: Total of all reporting groups
Arm/Group | Standard of Care Patients | TASKPEN Patients | Standard of Care Healthcare Providers | TASKPEN Healthcare Providers | Total
Number analyzed (Participants) | 634 | 456 | 20 | 8 | 1118
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: These data not collected for Healthcare Providers.
  years
    Participants: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    Participants | 46 [38 to 53] | 45 [38 to 52] |  |  | 45 [38 to 53]
Age, Customized [Count of Participants; unit: Participants] — Population: These data not collected for Healthcare Providers.
  Participants
    Participant age between 18-29: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    Participant age between 18-29 | 41 | 32 |  |  | 73
    Participant age between 30-44: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    Participant age between 30-44 | 246 | 185 |  |  | 431
    Participant age between 45-59: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    Participant age between 45-59 | 284 | 187 |  |  | 471
    Participant age between 60 and older: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    Participant age between 60 and older | 63 | 52 |  |  | 115
Sex: Female, Male [Count of Participants; unit: Participants] — Population: These data not collected for Healthcare Providers.
  Participants
    Participants: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    Participants: Female | 468 | 320 |  |  | 788
    Participants: Male | 166 | 136 |  |  | 302
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 634 | 456 | 20 | 8 | 1118
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 634 | 456 | 20 | 8 | 1118
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Zambia | 634 | 456 | 20 | 8 | 1118
Education [Count of Participants; unit: Participants] — Population: Data not collected for Healthcare Providers.
  Participants
    None: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    None | 45 | 55 |  |  | 100
    Primary: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    Primary | 276 | 238 |  |  | 514
    Secondary plus: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    Secondary plus | 313 | 163 |  |  | 476
Marital Status [Count of Participants; unit: Participants] — Population: Data not collected for Healthcare Providers.
  Participants
    Never married: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    Never married | 63 | 25 |  |  | 88
    Married or cohabitating: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    Married or cohabitating | 281 | 234 |  |  | 515
    Separated or Divorced or Widowed: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    Separated or Divorced or Widowed | 290 | 197 |  |  | 487
Body Mass Index (BMI) [Count of Participants; unit: Participants] — BMI was determined as follows: underweight is </= 18.49 Kg/m^2, healthy weight 18.5 to 24.99 Kg/m^2, overweight 25 to 29.99 Kg/m^2, and obese 30 or more Kg/m^2. Participants categorized as underweight, overweight, or obese were considered as having a worse outcome. Population: Data not collected for Healthcare Providers.
  Participants
    Underweight: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    Underweight | 53 | 41 |  |  | 94
    Healthy weight: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    Healthy weight | 257 | 246 |  |  | 503
    Overweight: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    Overweight | 178 | 107 |  |  | 285
    Obese: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    Obese | 146 | 56 |  |  | 202
    Missing data: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    Missing data | 0 | 6 |  |  | 6
Alcohol Consumption [Count of Participants; unit: Participants] — Population: Data not collected for Healthcare Providers.
  Participants
    Yes: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    Yes | 288 | 186 |  |  | 474
    No: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    No | 346 | 270 |  |  | 616
History of Hypertension [Count of Participants; unit: Participants] — Population: Data not collected for Healthcare Providers.
  Participants
    Yes: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    Yes | 151 | 129 |  |  | 280
    No: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    No | 483 | 327 |  |  | 810
History of Type II Diabetes [Count of Participants; unit: Participants] — Population: Data not collected for Healthcare Providers.
  Participants
    Yes: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    Yes | 23 | 10 |  |  | 33
    No: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    No | 603 | 445 |  |  | 1048
    Don't know: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    Don't know | 8 | 1 |  |  | 9
Time on ART [Count of Participants; unit: Participants] — Population: Data not collected for Healthcare Providers.
  Participants
    Less Than 5 Years: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    Less Than 5 Years | 139 | 87 |  |  | 226
    5-9 Years: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    5-9 Years | 141 | 111 |  |  | 252
    10 Years or more: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    10 Years or more | 354 | 258 |  |  | 612
History of Dyslipidemia [Count of Participants; unit: Participants] — Population: Data not collected for Healthcare Providers.
  Participants
    Yes: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    Yes | 1 | 2 |  |  | 3
    No: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    No | 631 | 454 |  |  | 1085
    Don't know: number analyzed (Participants) | 634 | 456 | 0 | 0 | 1090
    Don't know | 2 | 0 |  |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent of Participants With Dual HIV and Blood Pressure Control
Description: Measured by an HIV RNA level of <1000 copies per mL on the most recent measure and systolic blood pressure <140 mmHg and/or diasystolic blood pressure <90 mmHg. Dual control defined as HIV control (i.e., viral load <1,000 c/mL for those with a documented viral load + evidence of 6MMD for those with missing viral load) + Hypertension control (SBP<140 mmHg AND DBP<90 mmHg)
Time Frame: Baseline to 6 months
Population: Eleven patient participants with incomplete data were excluded.
Measure: Number; unit: percentage of participants
Groups:
- Standard of Care: During the control period, participants receive the current standard of care (SOC) in Zambia. Under the SOC in Zambian health facilities, the screening, diagnosis, and treatment of cardio-metabolic NCDs are generally unavailable in the clinical departments where most PLHIV seek and receive health services (i.e., ART and DSD clinics), and typically are only offered for hypertension in the general outpatient medical settings that provide urgent care-like services. Under the SOC, health worker capacity to diagnose and manage cardio-metabolic NCDs, including among non-physicians and community health workers, is severely limited and not protocolized like HIV services.
- TASKPEN: During the intervention period, participants receive TASKPEN intervention services.
  TASKPEN: The package of integrated HIV/NCD services:
  1. WHO PEN protocols, algorithm, & training materials adapted for Zambia
  2. Access to cardio-metabolic condition screening & laboratory monitoring
  3. Non communicable disease-focused electronic medical record module
  4. Integrated non-communicable/HIV care ("one stop shop" for services)
  5. Strengthened non-communicable disease (NCD) medication supply chain, including multi-month dispensing (MMD)
Arm/Group | Standard of Care | TASKPEN
Number analyzed (Participants) | 634 | 456
percentage of participants | 52 | 60

2. Secondary Outcome: Number of Clinics That Adopted the Intervention (Intervention Adoption)
Description: Adoption measured based on Reach Evaluation Adoption Implementation and Maintenance (RE-AIM) and Consolidated Framework for Implementation Research (CFIR) which are implementation-oriented and empirically supported frameworks for adapting, introducing, and evaluating evidence-based interventions in routine practice settings. The number of facilities initiating TASKPEN intervention integrated care at approximately 6 months after TASKPEN introduction.
Time Frame: 6 months
Measure: Count of Units; unit: Clinics
Units Other Than Participants: Clinics
Arm/Group | Standard of Care | TASKPEN
Number analyzed (Participants) | 636 | 465
Number analyzed (Clinics) | 2 | 2
Clinics | 1 | 1

3. Secondary Outcome: Number of Trained Healthcare Providers (Intervention Reach)
Description: Number of healthcare providers working at the pilot clinic antiretroviral therapy (ART), differentiated service delivery (DSD), and outpatient departments who were trained in the implementation of the TASKPEN intervention package.
Time Frame: During 2 weeks prior to initiation of TASKPEN
Population: The number of healthcare workers analyzed reflects the overall total number who were trained at the clinics and may include overlap from the Healthcare Providers enrolled to participate in the study survey.
Measure: Count of Participants; unit: Participants
Groups:
- Cluster 1 Healthcare Providers (George): 3 months without TASKPEN (Standard of Care (SOC)) and 6 months with TASKPEN.
  Training for Healthcare Providers was done at the time the clinic was switching from SOC to the TASKPEN intervention.
- Cluster 2 Healthcare Providers (Chilenje): 6 months without TASKPEN (Standard of Care (SOC)) and 3 months with TASKPEN.
  Training for Healthcare Providers was done at the time the clinic was switching from SOC to the TASKPEN intervention.
Arm/Group | Cluster 1 Healthcare Providers (George) | Cluster 2 Healthcare Providers (Chilenje)
Number analyzed (Participants) | 34 | 95
Participants | 29 | 60

4. Secondary Outcome: Changes in HIV Disease Control, as Measured by the Percent of Patient Participants With HIV RNA Suppression (Defined as <1,000 Copies/mL)
Description: Measured by the percent of patient participants with HIV RNA suppression (defined as <1,000 copies/mL)
Time Frame: Baseline to 6 months
Population: Data are reported for all patient participants with viral load test results available.
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care | TASKPEN
Number analyzed (Participants) | 542 | 406
percentage of participants | 85 | 89

5. Secondary Outcome: Change in Intervention Appropriateness
Description: The "Intervention appropriateness measure (IAM)" among healthcare providers. The minimum score is 1 and maximum is 5. Higher scores indicate greater appropriateness.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Healthcare Providers During Standard of Care: Healthcare Providers employed at the clinic overseeing patient participants during the control period (current standard of care (SOC)) in Zambia. Under the SOC in Zambian health facilities, the screening, diagnosis, and treatment of cardio-metabolic NCDs are generally unavailable in the clinical departments where most PLHIV seek and receive health services (i.e., ART and DSD clinics), and typically are only offered for hypertension in the general outpatient medical settings that provide urgent care-like services. Under the SOC, health worker capacity to diagnose and manage cardio-metabolic NCDs, including among non-physicians and community health workers, is severely limited and not protocolized like HIV services.
- Healthcare Providers During TASKPEN: Healthcare Providers employed at the clinic overseeing patient participants during the TASKPEN intervention service period.
  During the intervention period, patient participants receive TASKPEN intervention services.
  TASKPEN: The package of integrated HIV/NCD services:
  1. WHO PEN protocols, algorithm, & training materials adapted for Zambia
  2. Access to cardio-metabolic condition screening & laboratory monitoring
  3. Non communicable disease-focused electronic medical record module
  4. Integrated non-communicable/HIV care ("one stop shop" for services)
  5. Strengthened non-communicable disease (NCD) medication supply chain, including multi-month dispensing (MMD)
Arm/Group | Healthcare Providers During Standard of Care | Healthcare Providers During TASKPEN
Number analyzed (Participants) | 20 | 8
score on a scale | 4.69 (0.44) | 4.18 (0.39)

6. Secondary Outcome: Change in Intervention Acceptability
Description: Measured by the "Acceptability of Intervention measure (AIM)" among health care providers. The minimum score is 1 and maximum is 5. Higher scores indicate greater acceptability.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthcare Providers During Standard of Care | Healthcare Providers During TASKPEN
Number analyzed (Participants) | 20 | 8
score on a scale | 4.7 (0.44) | 4.34 (0.33)

7. Secondary Outcome: Change in Intervention Feasibility
Description: Measured by the "Feasibility of Intervention Measure (FIM)" among Healthcare providers. The minimum score is 1 and maximum is 5. Higher scores indicate greater feasibility.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthcare Providers During Standard of Care | Healthcare Providers During TASKPEN
Number analyzed (Participants) | 20 | 8
score on a scale | 4.66 (0.56) | 4.16 (0.44)

8. Secondary Outcome: Intervention Cost Per Patient
Description: Measured by cost per patient and reported in Zambian Kwacha. The analysis focused on the expenditures paid out of pocket for HIV and hypertension care. These data were collected from one site only (Chilenje).
Time Frame: 6 months
Population: These data were collected only at one study site. These data reflect out-of-pocket expenditures for participants living with HIV and at least one non-communicable disease co-morbidity.
Measure: Mean (Standard Error); unit: Kwacha (ZMW)
Groups:
- Standard of Care: 6 months without TASKPEN (Standard of Care (SOC)).
  During the control period, participants receive the current standard of care (SOC) in Zambia. Under the SOC in Zambian health facilities, the screening, diagnosis, and treatment of cardio-metabolic NCDs are generally unavailable in the clinical departments where most PLHIV seek and receive health services (i.e., ART and DSD clinics), and typically are only offered for hypertension in the general outpatient medical settings that provide urgent care-like services. Under the SOC, health worker capacity to diagnose and manage cardio-metabolic NCDs, including among non-physicians and community health workers, is severely limited and not protocolized like HIV services.
- TASKPEN: 3 months with TASKPEN
  During the intervention period, participants receive TASKPEN package of integrated HIV/NCD services:
  1. WHO PEN protocols, algorithm, & training materials adapted for Zambia
  2. Access to cardio-metabolic condition screening & laboratory monitoring
  3. Non communicable disease-focused electronic medical record module
  4. Integrated non-communicable/HIV care ("one stop shop" for services)
  5. Strengthened non-communicable disease (NCD) medication supply chain, including multi-month dispensing (MMD).
Arm/Group | Standard of Care | TASKPEN
Number analyzed (Participants) | 18 | 18
Kwacha (ZMW) | 352.53 (23.81) | 287.5 (101.02)

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through completion of each survey period, a combined total of 6 months.
Description: Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.0 November 2014. Adverse events were not collected for Healthcare Providers.
Arm/Group | Standard of Care | TASKPEN
All-Cause Mortality (participants affected / at risk) | 4/636 | 1/465
Serious Adverse Events (participants affected / at risk) | 0/636 | 0/465
Other Adverse Events (participants affected / at risk) | 158/636 | 222/465
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=636) | TASKPEN (N=465)
Hypertension (Cardiac disorders) | 143 (143) | 198 (198)
Out of Range Glucose (Endocrine disorders) | 15 (15) | 24 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/30/NCT05005130/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/30/NCT05005130/ICF_001.pdf